CLINICAL TRIAL: NCT01115751
Title: A Phase I Trial of Single-Agent LY2780301 in Patients With Advanced or Metastatic Cancer
Brief Title: A Study in Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13127; I4H-MC-JWAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-22; First posted 2010-05-04 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Metastases, Neoplasm
Keywords: Advanced Cancer; Metastatic Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2780301 (Experimental): Part A: daily dosing
  Part B (if determined as needed by pharmacokinetic, pharmacodynamic, and safety data): twice daily dosing
  Part C: Dose and frequency as determined by Parts A and B of the study.
  Interventions: Drug: LY2780301

INTERVENTIONS:
Drug: LY2780301 — Administered orally, daily for two 28-day cycles.
  Starting dose is 100mg. The dose will be subsequently increased to 200mg, 300mg, 400mg, 500mg, and 600mg if no dose limiting toxicity is observed at the prior dose levels. Patients who, in the opinion of the investigator, demonstrate clinical benefit may receive treatment beyond two cycles until disease progression.

SUMMARY:
Study JWAA is a multicenter, nonrandomized, open-label, dose-escalation Phase 1 study of oral LY2780301 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
JWAA will consist of the following treatment phases parts:

Part A - Dose escalation phase using a once-daily dosing schedule. Part B - Dose escalation phase using a twice-daily dosing schedule. Part C - Dose expansion phase using the maximum tolerated dose from either Part A or Part B.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic (including Non-Hodgkin's Lymphoma). The patient must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have failed to provide clinical benefit for their disease.
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or the Revised Response Criteria for Malignant Lymphoma.

Parts A and B: have measurable or nonmeasurable disease. Part C: have measurable disease.

* Have adequate organ function, including:

  * Hematologic: Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, platelets greater than or equal to 100 x 109/L, and hemoglobin greater than or equal to 8 g/dL. Transfusions are not allowed to reach 8 g/dL prior to enrollment.
  * Hepatic: Bilirubin less than or equal to 1.5 times upper limits of normal (ULN), alanine aminotransaminase (ALT), and aspartate aminotransaminase (AST) less than or equal to 2.5 times ULN. If the liver has tumor involvement, AST and ALT equaling less than or equal to 5 times ULN are acceptable.
  * Renal: Serum creatinine less than or equal to 1.5 times ULN or calculated creatinine clearance greater than 45 ml/mn.
* Have a performance status of less than or equal to 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued previous treatments for cancer and recovered from the acute effects of therapy: at least 28 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents. At the discretion of the investigator, hormone-refractory prostate cancer patients who are stable on gonadotropin-releasing hormone (GnRH) agonist therapy may have that treatment continued while they are enrolled in this study.

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication.
* Have serious preexisting medical conditions (left to the discretion of the investigator).
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required). Patients with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants, and their disease is asymptomatic and radiographically stable for at least 60 days.
* Have current acute or chronic leukemia.
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).
* Have a second primary malignancy that in the judgment of the investigator and sponsor may affect the interpretation of results.
* Have QTc interval of >470 msec on screening electrocardiogram(ECG).
* Treatment with a strong CYP3A4 substrate with narrow therapeutic range, strong inhibitor, or inducer.
* Have history of pituitary adenoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Recommended dose for Phase 2 Studies | Baseline to study completion

SECONDARY OUTCOMES:
Clinically significant effects | Baseline to study completion
Pharmacokinetics, area under the concentration-time curve | Baseline, Days 1, 2, 8, 15, and 22 of Cycle 1, Day 1 of Cycle 2
Best overall response (CR+PR+SD) | Baseline to measured disease progression. Tumor assessments are performed every 2 cycles until disease progression and during post-study follow-up period.
Progression-free survival | Baseline to measured disease progression or death. Tumor assessments are performed every 2 cycles until disease progression and during post-study follow-up period.
Duration of response | Time of response to disease progression or death. Tumor assessments are performed every 2 cycles until disease progression and during post-study follow-up period.
Pharmacokinetics, maximum concentration (Cmax) | Baseline, Days 1, 2, 8, 15, and 22 of Cycle 1, Day 1 of Cycle 2

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid